CLINICAL TRIAL: NCT07204652
Title: Detection of Phosphorylated Alpha-synuclein Through Routine Colonoscopy to Diagnose Parkinson's Disease and Related Disorders
Brief Title: Colonoscopic Detection of Phosphorylated Alpha-synuclein for Parkinson's Diagnosis
Acronym: Syn-G
Status: Recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: OHSU IRB # 27731
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson; Parkinson's Disease and Parkinsonism; Parkinson Disease
Keywords: Parkinson; Parkinson's Disease; Parkinson disease; Parkinson Disease (Disorder)
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
The goal of this observational study is to learn whether tissue samples taken from the colon during routine colonoscopy can detect signs of Parkinson's disease. The main question it aims to answer is:

Can doctors find a protein called alpha-synuclein in colon tissue samples from people with Parkinson's disease?

Currently, Parkinson's disease is diagnosed by observing symptoms like tremors and movement problems, but by then the disease has already progressed significantly. Earlier detection could help doctors start treatment sooner.

DETAILED DESCRIPTION:
Brief Summary

What is this study about? This study is testing whether doctors can detect signs of Parkinson's disease by taking small tissue samples from the colon during a routine colonoscopy. Researchers want to see if they can find a specific protein called alpha-synuclein that builds up in people with Parkinson's disease.

Why is this study important? Currently, Parkinson's disease is diagnosed mainly by observing symptoms like tremors and movement problems. However, by the time these symptoms appear, the disease has already progressed significantly. Finding a way to detect the disease earlier could help doctors start treatment sooner and potentially slow down the disease.

Who can participate?

* Adults between 40-99 years old
* People who have already been diagnosed with Parkinson's disease
* People who are already scheduled to have a routine colonoscopy for colon cancer screening or other medical reasons

What happens during the study? **Before the colonoscopy:**

* Participants will complete questionnaires about their Parkinson's symptoms, sleep, and thinking abilities
* They will take a brief smell test
* They will collect a stool sample at home using a provided kit

**During the colonoscopy:**

* The colonoscopy procedure remains exactly the same as planned
* Doctors will take 4 additional small tissue samples (2 from each side of the colon)
* This adds only about 2 minutes to the procedure

**After the colonoscopy:**

* No additional visits are required
* The tissue samples will be tested for the alpha-synuclein protein
* Participants will not receive individual test results

What are the risks?

The main risks are the same as any routine colonoscopy, including:

* Discomfort during the procedure
* Very rare complications like bleeding or bowel perforation
* Small risk of infection
* Possible breach of medical privacy (researchers take steps to protect this)

What are the benefits?

* Participants help advance research that could lead to earlier detection of Parkinson's disease
* This could eventually help future patients get diagnosed and treated sooner
* There are no direct medical benefits to participants

How many people will be in this study? 20 people with Parkinson's disease will participate in this study at Oregon Health & Science University (OHSU).

How long does participation take?

* One screening visit before the colonoscopy (about 1-2 hours)
* The colonoscopy procedure (same length as normally planned)
* Collecting a stool sample at home (one time)

This research is sponsored by CND Life Sciences and conducted at OHSU.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40 to 99 years of age
* Patients with a confirmed clinical diagnosis of Parkinson's disease by UKPDS Brain Bank Criteria
* Patients who have agreed to undergo a routine colonoscopy as part of their surveillance for colon cancer or exclusion of other gastrointestinal diseases

Exclusion Criteria:

* Use of anticoagulants (Plavix 75 mg or aspirin up to 325 mg alone is allowed)
* History of colon cancer
* Recent gastrointestinal illness or surgical procedures
* Pregnant or planning to become pregnant before the scheduled colonoscopy
* Significant cognitive impairment, as determined by study investigators
* Decisionally impaired adults who cannot express understanding that this study is voluntary and for research purposes

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinically confirmed Parkinson's disease who are undergoing routine colonoscopies for standard medical care. Participants must be able to provide informed consent and understand that participation is voluntary and for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Detection of phosphorylated alpha-synuclein in colon tissue samples | At time of colonoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Delaram Safarpour, MD, MSCE, FAAN, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States